CLINICAL TRIAL: NCT00289679
Title: Cytokine Profile and Metal Ion Concentrations at Patients Undergoing a Revision THR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frederiksberg University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: kf 01059/04
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2007-07

CONDITIONS: Hip Revision

INTERVENTIONS:
Device: Hip prosthesis revision

SUMMARY:
To evaluate the concentration of cytokines and metal ions in blod samples and biopsies from patients undergoing a hip revision.

ELIGIBILITY:
Inclusion Criteria:

* THR revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: arne borgwardt, md, Principal Investigator — Frederiksberg University Hospital
Locations (1):
- Frederiksberg University Hospital, Frederiksberg, Frederiksberg, Denmark